CLINICAL TRIAL: NCT06880718
Title: Injectable Buprenorphine During Transition Out of Prison: a Partially Randomized Preference Pilot Trial
Brief Title: Injectable Buprenorphine in Prison: a Preference Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Justin Berk, Assistant Professor, Lifespan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2210402; K23DA055695 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder; Incarceration; Medications for Opioid Use Disorder; Buprenorphine
Keywords: opioid use disorder; incarceration; prison; long-acting injectable; buprenorphine; XR-B
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sublocade (Active Comparator): Participants receive Sublocade-branded injectable buprenorphine.
  Interventions: Drug: Sublocade
- Brixadi (Active Comparator): Participants receive Brixadi-branded injectable buprenorphine.
  Interventions: Drug: Brixadi (Injectable Buprenorphine)

INTERVENTIONS:
Drug: Brixadi (Injectable Buprenorphine) — Brixadi comes in several doses and can be administered on a weekly or monthly basis. For clinical reasons (i.e., each patient will already be on a stable dose of MOUD in a setting without significant illicit opioid use), the monthly injection will be used. The approximately equivalent to the 300mg Sublocade dose is 96mg of Brixadi. The maximum dose is 128mg. Brixadi can be administered in the abdomen, buttocks, or triceps. Participants in the Brixadi treatment arm will be given one or more Brixadi injections each month prior to release from prison and each month after release. They can continue to receive the medication after the conclusion of the trial. Brixadi is covered by most Medicaid health insurances in the state of Rhode Island.
  Other Names: CAM2308; Buvidal
  Arms: Brixadi
Drug: Sublocade — Sublocade is a 100mg or 300mg pre-mixed subcutaneous injectable formulation to be administered monthly. Participants in the Sublocade treatment arm will be given monthly Sublocade injections, as clinically indicated, each month prior to release from prison and each month after release. They can continue to receive the medication after the conclusion of the trial. Sublocade is covered by most Medicaid health insurances in the state of Rhode Island. The standard dosing schedule is two months of 300mg followed by monthly 100mg injections. To maximize real-world generalizability, the medication dosing will be determined by clinical indication of the provider who will have the flexibility to provide medication dosing based on their clinical acumen and/or shared decision-making.
  Arms: Sublocade

SUMMARY:
The goal of this pilot trial is to compare two branded extended-release buprenorphine (XR-B) formulations (Sublocade vs. Brixadi) to explore how they improve treatment retention after release from prison among incarcerated individuals with opioid use disorder (OUD) who are transitioning back into the community.

The main question it aims to answer are:

How do Sublocade and Brixadi compare in terms of feasibility, acceptability, and effectiveness? Does giving people a choice of medication affect how well they stay in treatment?

Using a partially randomized preference trial approach, there will be a comparison between participants who choose their XR-B formulation to those who are randomly assigned to see if patient preference influences treatment outcomes. The trial is a hybrid implementation-effectiveness trial.

Participants will:

* Choose which medication they prefer or be randomly assigned if they don't have a preference.
* Receive monthly injections of either Sublocade or Brixadi before and after release from prison.
* Complete surveys and clinical assessments on treatment experience and acceptability.
* Be monitored for treatment retention, opioid use, and adverse events for six months post-release.

Researchers will compare the two treatments to see which one works better for people leaving prison and if allowing people to choose their treatment improves results.

DETAILED DESCRIPTION:
This study is a pilot hybrid effectiveness-implementation trial using a partially randomized preference trial (PRPT) design to evaluate two formulations of extended-release buprenorphine (XR-B)-Sublocade and Brixadi-for the treatment of opioid use disorder (OUD) in individuals transitioning from prison to the community. The study is being conducted in collaboration with the Rhode Island Department of Corrections (RIDOC) to assess treatment retention, feasibility, and acceptability and other implementation outcomes in a carceral setting.

STUDY OBJECTIVES As a hybrid trial, the study will assess effectiveness and implementation outcomes. The primary objective of this study is to compare effectiveness (post-release treatment retention) among participants who receive Sublocade or Brixadi before and after release from prison. The study also aims to evaluate the impact of patient preference on treatment outcomes, including differences in retention between those who choose their treatment and those who are randomized. The study will also assess implementation outcomes including feasibility, acceptability, and fidelity.

STUDY DESIGN This is a pilot hybrid effectiveness-implementation trial that incorporates a partially randomized preference trial (PRPT) design.

Participants with a clear preference for either Sublocade or Brixadi will receive their preferred treatment. Participants with no strong preference will be randomized 1:1 using a stratified block randomization approach, stratified by gender, with blocks of four. Randomization assignments will be concealed using opaque sealed envelopes. The study is open-label, meaning both participants and study staff will be aware of treatment assignments. Given the preference-based design, blinding is not feasible.

STUDY SETTING The study will recruit participants from RIDOC, which has a long-standing MOUD program. Eligible participants are incarcerated individuals with upcoming release dates that express interest in XR-B and have no contraindications to treatment.

INTERVENTION Participants will receive either Sublocade or Brixadi based on their assignment. Interventions will be provided monthly. Participants are allowed to change treatments or discontinue any time.

OUTCOME MEASURES

The study will assess implementation, service, and client outcomes based on the Proctor et al. framework:

1. Implementation Outcomes (acceptability, feasibility, appropriateness, fidelity) Acceptability: Initial treatment preferences, in-facility retention, and the Acceptability of Intervention Measure (AIM).

   Feasibility: Feasibility of Intervention Measure (FIM) and study enrollment rates.

   Appropriateness: Intervention Appropriateness Measure (IAM). Fidelity: Proportion of XR-B doses administered within the appropriate dosing window (26-35 days).
2. Service Outcomes (effectiveness, safety, equity) Effectiveness: Post-release retention in MOUD treatment Safety: Incidence of adverse events associated with XR-B administration.
3. Client Outcomes (satisfaction, function, symptomatology) Treatment Satisfaction: Modified Treatment Satisfaction Questionnaire (TSQM-9). Opioid Use: Self-reported opioid use and urine toxicology screens (with missing tests assumed positive).

Health Service Utilization: Emergency department visits and hospitalizations (tracked via electronic health records).

Cravings: Opioid Craving Visual Analog Scale (OC-VAS).

SAMPLE SIZE This is a pilot study with a target enrollment of 60 participants (30 per treatment arm).

DATA COLLECTION Data Sources: Data will be collected through self-reported surveys, clinical records, urine toxicology tests, and statewide administrative databases (including the Rhode Island Prescription Drug Monitoring Program).

Data Security: All identifiable information will be stored in a secure, HIPAA-compliant system with restricted access.

STATISTICAL ANALYSIS PLAN Primary Analysis: Logistic regression will be used to compare treatment retention across study arms.

Secondary Analyses: Feasibility, acceptability, and safety outcomes will be analyzed using ordinal logistic regression (e.g., AIM, FIM, IAM). Kaplan-Meier survival curves will assess time-to-treatment discontinuation. Generalized estimating equations (GEE) will be used to model repeated measures outcomes such as opioid cravings and treatment satisfaction over time. Differences in treatment satisfaction and opioid use will be analyzed using linear regression for continuous variables and logistic regression for binary variables.

Sensitivity Analysis: Sensitivity analyses will include intent-to-treat (ITT), per-protocol (PP), and modified intent-to-treat (mITT) approaches. ITT analysis will include all randomized participants in their assigned groups, regardless of treatment adherence. PP analysis will focus on participants who complete at least two months of XR-B post-release to assess effectiveness among those who adhere to treatment. The mITT analysis will exclude participants who become ineligible due to changes in release dates post-enrollment to better estimate true treatment effects. Multiple imputation will be used for missing data, and additional sensitivity analyses will assess the robustness of findings across different assumptions regarding missingness.

SAFETY MONITORING AND ADVERSE EVENTS Adverse events (AEs) and serious adverse events (SAEs) will be monitored using the Systematic Assessment for Treatment Emergent Events (SAFTEE) framework. A Data and Safety Monitoring Board (DSMB) will oversee study progress and participant safety. All unanticipated problems, protocol deviations, and safety concerns will be reported to the Brown University Health IRB and RIDOC Medical Review Board.

LIMITATIONS As a pilot study, this study is not powered to detect small differences in effectiveness. Findings may not generalize beyond Rhode Island's correctional system. Findings will inform a larger, multi-site hybrid trial evaluating XR-B formulations in diverse correctional settings.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years of age and incarcerated in the RIDOC facility,
2. be currently diagnosed with OUD and enrolled in the RIDOC MOUD program,
3. have an expected release date within 120 days of study enrollment,
4. have an interest in XR-B and
5. be English speaking

Exclusion Criteria:

1. individuals who are pregnant or planning conception,
2. diagnosed with a severe or acute medical or psychiatric disability preventing safe study participation or making follow-up unlikely,
3. have a release date within 21 days of initiation, or
4. have previously had an allergy to buprenorphine. Post-enrollment exclusion will include individuals if there is a change in release date beyond the 120 days and therefore no longer meet original inclusion criteria. These individuals would return to usual MOUD care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Preliminary Effectiveness | 3 months post-release
  Preliminary Effectiveness will be measured through rates of community treatment continuation post-release. Outpatient treatment engagement over the first three months post-release will be assessed using study records of CPC Recovery Clinic follow-up appointments. For patients that do not follow at the CPC Recovery Clinic, statewide administrative data from the Rhode Island Prescription Drug Monitoring Program (PDMP) database covering community pharmacy fills of buprenorphine products will be used to supplement treatment retention outcomes. PDMP data will also be used to track community treatment continuation for all participants from three to six months post-release. Participants will be logged as continuing buprenorphine treatment at each month if: (1) CPC Recovery Clinic records show that they were present at their scheduled follow-up visit, or (2) the PDMP indicates that they continued treatment elsewhere and have not had a gap of more than 30 days in dispensed medication.
Implementation Outcomes: Acceptability | Baseline, Immediately after the intervention
  Acceptability will be measured through initial patient preference, in-facility treatment retention, and the validated Acceptability of Intervention Measure (AIM).
  The Acceptability of Intervention Measure (AIM) assesses the extent to which an intervention is perceived as satisfactory or agreeable by stakeholders. Scores are calculated using a 5-point Likert scale, where 1 = Completely Disagree and 5 = Completely Agree. The minimum possible score is 1, and the maximum possible score is 5. Higher scores indicate greater acceptability of the intervention.
Implementation Outcomes: Feasibility | Baseline, Immediately after the intervention
  Feasibility will be measured by the validated Feasibility of Intervention Measure (FIM) and enrollment rates.
  The Feasibility of Intervention Measure (FIM) evaluates the degree to which an intervention can be successfully used or implemented within a given setting. Scores are calculated using a 5-point Likert scale, where 1 = Completely Disagree and 5 = Completely Agree. The minimum possible score is 1, and the maximum possible score is 5. Higher scores indicate greater feasibility of implementing the intervention.
Implementation Outcomes: Appropriateness | Baseline, Immediately after the intervention
  Appropriateness will be measured by the validated Intervention Appropriateness Measure (IAM).
  The Appropriateness of Intervention Measure (IAM) measures how well an intervention fits with the setting, needs, or problem it is intended to address. Scores are calculated using a 5-point Likert scale, where 1 = Completely Disagree and 5 = Completely Agree. The minimum possible score is 1, and the maximum possible score is 5. Higher scores indicate greater perceived appropriateness of the intervention.
Implementation Outcomes: Fidelity | Baseline, Immediately after the intervention
  Fidelity will be measured by the proportion of doses administered within the 26-35 day range of appropriate dosing cadence.

SECONDARY OUTCOMES:
Client Outcomes: Satisfaction | During the intervention
  Treatment Satisfaction will be assessed using a modified version of the previously validated Treatment Satisfaction Questionnaire for Medication (TSQM-9) after each in-facility injection.
  TSQM scoring is by domain and each domain score is computed by summing the individual TSQM items in each domain and then transforming the composite score into a value ranging from 0 to 100, 100 as highly satisfied.
Client Outcomes: Function - Healthcare Utilization | During the intervention
  Healthcare utilization will be assessed using emergency department or hospital visits will be tracked using Rhode Island Hospital CPC Recovery Clinic Electronic Medical Record data.
Client Outcomes: Function - Recidivism | During the intervention, 3 months after the intervention
  Reincarceration will be tracked using RIDOC administrative data identifying return to jail or prison.
Client Outcomes: Treatment Satisfaction | During the intervention
  Treatment Satisfaction will be assessed using a modified version of the previously validated Treatment Satisfaction Questionnaire for Medication (TSQM-9) after each in-facility injection.
Client Outcomes: Function - Return to Use | During the intervention
  Illicit opioid abstinence will be assessed through urine toxicology screening at each CPC Recovery Clinic follow-up appointment.

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and study results have been published, de-identified data will be made available to other qualified researchers upon request. Each data request will be evaluated by the PI to ensure that it meets reasonable standards of scientific integrity. The researchers have carefully selected standardized and widely-used assessments to promote data sharing and integration into larger databases and to allow other researchers the ability to analyze the data, including by conducting meta-analyses. The researchers will submit primary results for publication by the end of the project period and will have final de-identified datasets available within six months of the end of the project period.
Supporting Information: Study Protocol